CLINICAL TRIAL: NCT01688856
Title: Optimizing Contralaterally Controlled FES for Acute Upper Limb Hemiplegia
Brief Title: Contralaterally Controlled FES of Arm & Hand for Subacute Stroke Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MetroHealth Medical Center (Other)
Collaborators: Case Western Reserve University (Other); National Institutes of Health (NIH) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Jayme Knutson, Assistant Professor, Physical Medicine and Rehabilitation, MetroHealth Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB12-00493; R01HD068588 (NIH)
Record Dates: First submitted 2012-09-17; First posted 2012-09-20 (Estimated); Results first posted 2020-01-09 (Actual); Last update posted 2020-01-09 (Actual); Status verified 2020-01

CONDITIONS: Stroke; Hemiparesis; Hemiplegia
Keywords: hand; arm; stroke; hemiplegia; electrical stimulation; recovery; rehabilitation
MeSH Terms: conditions — Stroke; Paresis; Hemiplegia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm+Hand CCFES (Experimental): Uses an electrical stimulator that opens the paretic hand and extends the paretic elbow in response to and with an intensity proportional to movement of the contralateral arm and hand. The treatment dose will be approximately 2 hrs per day of self-administered stimulation-mediated exercise at home plus 70 min of functional task practice twice a week in the laboratory for 12 weeks.
  Interventions: Device: Electrical Stimulator
- Hand CCFES (Experimental): Uses an electrical stimulator that opens the paretic hand in response to and with an intensity proportional to movement of the contralateral hand. The treatment dose will be approximately 2 hrs per day of self-administered stimulation-mediated exercise at home plus 70 min of functional task practice twice a week in the laboratory for 12 weeks.
  Interventions: Device: Electrical Stimulator
- Arm+Hand Cyclic NMES (Active Comparator): Uses an electrical stimulator that delivers stimulation to open the hand and extend the elbow repeatedly with preprogrammed timing and intensity. The treatment dose will be approximately 2 hrs per day of self-administered stimulation-mediated exercise at home plus 70 min of functional task practice twice a week in the laboratory for 12 weeks.
  Interventions: Device: Electrical Stimulator

INTERVENTIONS:
Device: Electrical Stimulator — The 12-week treatment period consists of two components:
  1. Therapist-guided task practice performed 70 minutes twice a week in the research laboratory. If Arm+Hand CCFES or Hand CCFES, the stimulator is used during task practice.
  2. Self-administered muscle stimulation exercise performed 10 sessions per week at home using the device. If Arm+Hand CCFES or Hand CCFES, each session is 46 minutes. If Arm+Hand Cyclic NMES, each session is 60 minutes.

SUMMARY:
Impaired arm and hand function is one of the most disabling and most common consequences of stroke. The Investigators have developed Contralaterally Controlled Functional Electrical Stimulation (CCFES), an innovative neuromuscular electrical stimulation (NMES) treatment for improving the recovery of hand function after stroke. The purpose of this study is to maximize the treatment effect of CCFES by adding stimulated elbow extension. The specific aims and hypotheses are as follows:

AIM 1: Estimate the effect of Arm+Hand CCFES on upper limb motor impairment and activity limitation.

Hypothesis 1: Stroke survivors treated with Arm+Hand CCFES have better outcomes on upper limb impairment and activity limitation measures than those treated with dose-matched Arm+Hand Cyclic NMES.

AIM 2: Estimate the effect of adding stimulated elbow extension to Hand CCFES.

Hypothesis 2: Stroke survivors treated with Arm+Hand CCFES will have greater reductions in upper limb impairment and activity limitation than those treated with Hand CCFES.

AIM 3: Describe the relationship between treatment effect and time elapsed between stroke onset and start of treatment.

Hypothesis 3: Patients who start Arm+Hand CCFES sooner after their stroke achieve better outcomes.

DETAILED DESCRIPTION:
Loss of arm and hand function is a severely disabling condition that occurs in nearly 75% of the estimated 795,000 Americans who have a new or recurrent stroke each year [Roger 2011]. Upper limb impairment is often characterized by inability to extend the elbow and open the hand. The hope of regaining lost motor function after stroke has been fueled in recent years by the development of new rehabilitation therapies and devices that are aimed at promoting the brain's capacity to reorganize after injury in such a way that restores motor control of paretic limbs [Nudo 2001]. The Investigators' long-term objective is to develop stroke rehabilitation treatments for the hemiparetic upper limb that are optimized for effectiveness, applicability, and deployability.

The primary objective of this project is to estimate the effect of Arm+Hand Contralaterally Controlled Functional Electrical Stimulation (CCFES) in reducing upper limb motor impairment and activity limitation in subacute hemiplegia. CCFES is a treatment aimed at improving recovery of volitional motor function in stroke survivors [Knutson 2007; Knutson 2009; Knutson 2010]. Hand CCFES activates finger and thumb extensors with an intensity of electrical stimulation that is proportional to the degree of opening of the contralateral unimpaired hand wearing an instrumented glove. Thus, volitional opening of the nonparetic hand produces stimulated opening of the paretic hand. The Hand CCFES system enables stroke patients to use their impaired hand to practice functional tasks in therapy sessions. CCFES incorporates the following features considered to be important to motor recovery and promoting neuroplasticity: synchronization of motor intent with motor execution of paretic hand opening [Rushton 2003; Kimberley 2004], bilateral symmetric movement [Luft 2004], intensive repetitive hand opening exercises [Lang 2009], and the practice of functional tasks [Nudo 2003]. In a pilot case series study of patients with chronic (> 6 months) post-stroke hemiplegia, all 6 participants experienced some reduction of upper limb motor impairment after several weeks of Hand CCFES [Knutson 2007; Knutson 2009]. The results of a Phase I randomized clinical trial (RCT) of Hand CCFES in 21 patients with subacute (≤ 6 months) hemiplegia suggested that Hand CCFES may be superior to cyclic neuromuscular electrical stimulation (NMES) in reducing upper extremity impairment and activity limitation [Knutson 2011].

In this study, added to the Hand CCFES treatment is stimulated elbow extension controlled by the contralateral elbow. This "next generation" CCFES treatment is called Arm+Hand CCFES. Arm+Hand CCFES therapy is intended to strengthen and improve the motor control of the proximal upper limb as well as the hand, to improve simultaneous reaching and hand opening, a functionally critical movement pattern that is often prevented by paresis and post-stroke flexor synergies. The secondary objective of this project is to evaluate the effect of adding elbow extensor stimulation to the Hand CCFES treatment.

Stroke survivors who are ≤ 2 years post-stroke with upper limb hemiplegia will be randomly assigned to receive 12 weeks of either Arm+Hand CCFES (stimulates elbow extension and hand opening), Hand CCFES (stimulates hand opening), or Arm+Hand Cyclic NMES (stimulates elbow extension and hand opening but with pre-set timing and intensity, i.e., not intention-driven), plus lab-based therapist-guided task practice. Upper limb impairment and activity limitation will be assessed at baseline, 6, 12, 20, 28, and 36 weeks.

This is the first randomized controlled trial of Arm+Hand CCFES in subacute upper extremity hemiplegia. Ultimately, the information learned in this study will serve to accelerate the development of a new treatment for reducing post-stroke disability.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 21 and ≤ 80
* ≤ 2 years of first clinical hemorrhagic or nonhemorrhagic stroke
* Skin intact on hemiparetic arm and hand
* Able to follow 3-stage commands
* Able to recall 2 of 3 items after 30 minutes
* Medically stable
* Finger extensor paresis indicated by a score of ≤ 4 out of 5 on the manual muscle test (Medical Research Council scale)
* Adequate movement of shoulder and elbow to position the paretic hand in the workspace for table-top task practice
* Caregiver available to assist with device daily - OR - able to independently don elbow cuff on unaffected arm
* Full volitional elbow extension/flexion and hand opening/closing of unaffected limb
* Upper extremity hand section of Upper Extremity Fugl-Meyer (UEFM)≥ 1 AND ≤ 11/14
* Unable to simultaneously fully extend the elbow and fully open the hand toward tabletop object with arm unsupported (i.e. cannot voluntarily achieve the maximum passive range of motion (PROM) available)
* Functional PROM (minimal resistance) at shoulder, elbow, wrist, and hand simultaneously on affected side (i.e., there exists enough PROM to reach and acquire table-top objects).
* Able to hear and respond to stimulator cues
* While relaxed, surface NMES of finger extensors and thumb extensors and/or abductors produces a functional degree of hand opening without pain.
* While relaxed with the forearm supported with a mobile arm support, surface NMES of elbow extensors (triceps) produces functional elbow extension without pain.
* Patient must be able to sit unassisted in an armless straight-back chair for the duration of the screening portion of the eligibility assessment.

Exclusion Criteria:

* Co-existing neurological condition other than prior stroke involving the hemiparetic upper limb (e.g., peripheral nerve injury, Parkinson's Disease, Spinal Cord Injury, Traumatic Brain Injury, Multiple Sclerosis).
* Severely impaired cognition and communication
* Uncontrolled seizure disorder
* History of cardiac arrhythmias with hemodynamic instability
* Cardiac pacemaker or other implanted electronic device
* Pregnant
* IM Botox injections in any UE muscle in the last 3 months
* Insensate arm, forearm, or hand
* Uncompensated hemi-neglect (extinguishing to double simultaneous stimulation)
* Severe shoulder or hand pain
* Severe depression on Beck Depression Inventory (BDI) (score>=13 on BDI-fast screen)

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2018-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jayme S. Knutson, PhD, Principal Investigator — MetroHealth Medical Center
Locations (1):
- MetroHealth Medical Center, Cleveland, Ohio, United States

REFERENCES:
- [Background] Nudo RJ, Plautz EJ, Frost SB. Role of adaptive plasticity in recovery of function after damage to motor cortex. Muscle Nerve. 2001 Aug;24(8):1000-19. doi: 10.1002/mus.1104. PMID 11439375
- [Background] Knutson JS, Harley MY, Hisel TZ, Chae J. Improving hand function in stroke survivors: a pilot study of contralaterally controlled functional electric stimulation in chronic hemiplegia. Arch Phys Med Rehabil. 2007 Apr;88(4):513-20. doi: 10.1016/j.apmr.2007.01.003. PMID 17398254
- [Background] Knutson JS, Hisel TZ, Harley MY, Chae J. A novel functional electrical stimulation treatment for recovery of hand function in hemiplegia: 12-week pilot study. Neurorehabil Neural Repair. 2009 Jan;23(1):17-25. doi: 10.1177/1545968308317577. Epub 2008 Sep 23. PMID 18812432
- [Background] Knutson JS, Chae J. A novel neuromuscular electrical stimulation treatment for recovery of ankle dorsiflexion in chronic hemiplegia: a case series pilot study. Am J Phys Med Rehabil. 2010 Aug;89(8):672-82. doi: 10.1097/PHM.0b013e3181e29bd7. PMID 20531158
- [Background] Kimberley TJ, Lewis SM, Auerbach EJ, Dorsey LL, Lojovich JM, Carey JR. Electrical stimulation driving functional improvements and cortical changes in subjects with stroke. Exp Brain Res. 2004 Feb;154(4):450-60. doi: 10.1007/s00221-003-1695-y. Epub 2003 Nov 15. PMID 14618287
- [Background] Rushton DN. Functional electrical stimulation and rehabilitation--an hypothesis. Med Eng Phys. 2003 Jan;25(1):75-8. doi: 10.1016/s1350-4533(02)00040-1. PMID 12485788
- [Background] Luft AR, McCombe-Waller S, Whitall J, Forrester LW, Macko R, Sorkin JD, Schulz JB, Goldberg AP, Hanley DF. Repetitive bilateral arm training and motor cortex activation in chronic stroke: a randomized controlled trial. JAMA. 2004 Oct 20;292(15):1853-61. doi: 10.1001/jama.292.15.1853. PMID 15494583
- [Background] Lang CE, Macdonald JR, Reisman DS, Boyd L, Jacobson Kimberley T, Schindler-Ivens SM, Hornby TG, Ross SA, Scheets PL. Observation of amounts of movement practice provided during stroke rehabilitation. Arch Phys Med Rehabil. 2009 Oct;90(10):1692-8. doi: 10.1016/j.apmr.2009.04.005. PMID 19801058
- [Background] Nudo RJ. Adaptive plasticity in motor cortex: implications for rehabilitation after brain injury. J Rehabil Med. 2003 May;(41 Suppl):7-10. doi: 10.1080/16501960310010070. PMID 12817650
- [Background] Knutson JS, Harley MY, Hisel TZ, Hogan SD, Maloney MM, Chae J. Contralaterally controlled functional electrical stimulation for upper extremity hemiplegia: an early-phase randomized clinical trial in subacute stroke patients. Neurorehabil Neural Repair. 2012 Mar-Apr;26(3):239-46. doi: 10.1177/1545968311419301. Epub 2011 Aug 29. PMID 21875892
- [Background] Roger VL, Go AS, Lloyd-Jones DM, Adams RJ, Berry JD, Brown TM, Carnethon MR, Dai S, de Simone G, Ford ES, Fox CS, Fullerton HJ, Gillespie C, Greenlund KJ, Hailpern SM, Heit JA, Ho PM, Howard VJ, Kissela BM, Kittner SJ, Lackland DT, Lichtman JH, Lisabeth LD, Makuc DM, Marcus GM, Marelli A, Matchar DB, McDermott MM, Meigs JB, Moy CS, Mozaffarian D, Mussolino ME, Nichol G, Paynter NP, Rosamond WD, Sorlie PD, Stafford RS, Turan TN, Turner MB, Wong ND, Wylie-Rosett J; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Heart disease and stroke statistics--2011 update: a report from the American Heart Association. Circulation. 2011 Feb 1;123(4):e18-e209. doi: 10.1161/CIR.0b013e3182009701. Epub 2010 Dec 15. PMID 21160056
- [Derived] Knutson JS, Friedl AS, Hansen KM, Hisel TZ, Harley MY. Convergent Validity and Responsiveness of the SULCS. Arch Phys Med Rehabil. 2019 Jan;100(1):140-143.e1. doi: 10.1016/j.apmr.2018.07.433. Epub 2018 Aug 24. PMID 30148996
- See also: Cleveland FES Center — http://fescenter.org/index.php

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm+Hand CCFES: Uses an electrical stimulator that opens the paretic hand and extends the paretic elbow in response to and with an intensity proportional to movement of the contralateral arm and hand.
  Electrical stimulator: The 12-week treatment period consists of two components:
  1. Therapist-guided CCFES-mediated task practice performed 70 minutes twice a week in the research laboratory.
  2. Self-administered hand opening exercise performed 10 sessions per week at home using the device. 46 min/session.
- Hand CCFES: Uses an electrical stimulator that opens the paretic hand in response to and with an intensity proportional to movement of the contralateral hand.
  Electrical stimulator: The 12-week treatment period consists of two components:
  1. Therapist-guided CCFES-mediated task practice performed 70 minutes twice a week in the research laboratory.
  2. Self-administered hand opening exercise performed 10 sessions per week at home using the device. 46 min/session.
- Arm+Hand Cyclic NMES: Uses an electrical stimulator that delivers stimulation to open the hand and extend the elbow repeatedly with preprogrammed timing and intensity.
  Electrical stimulator: The 12-week treatment period consists of two components:
  1. Therapist-guided task practice performed 70 minutes twice a week in the research laboratory. (Stimulator not used during these sessions. To ensure that all 3 groups receive an equivalent dose of stimulation, this group has slightly lengthened self-administered hand opening exercise sessions at home.)
  2. Self-administered hand opening exercise performed 10 sessions per week at home using the device. 60 min/session.
Period: Overall Study
Arm/Group | Arm+Hand CCFES | Hand CCFES | Arm+Hand Cyclic NMES
Started | 28 | 28 | 11
Completed | 21 | 24 | 8
Not Completed | 7 | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm+Hand CCFES | Hand CCFES | Arm+Hand Cyclic NMES | Total
Number analyzed (Participants) | 28 | 28 | 11 | 67
Age, Continuous [Mean (Standard Deviation); unit: years] | 54 (12.6) | 60 (11.5) | 61 (12.5) | 58 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 7 | 8 | 24
  Male | 19 | 21 | 3 | 43
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 13 | 7 | 2 | 22
  White | 13 | 19 | 9 | 41
  Other | 2 | 2 | 0 | 4

OUTCOME MEASURES:

1. Primary Outcome: Change in Box and Block Test (BBT) Score at 6 Months Post-Treatment
Description: The BBT counts how many blocks a participant can pick up, move over a barrier, and release in 60 seconds. Higher scores mean a better outcome.
Time Frame: 2 timepoints: prior to treatment, 6 months post-treatment
Measure: Least Squares Mean (95% Confidence Interval); unit: blocks
Arm/Group | Arm+Hand CCFES | Hand CCFES | Arm+Hand Cyclic NMES
Number analyzed (Participants) | 21 | 24 | 8
blocks | 13.5 [6.4 to 20.6] | 12.6 [7.4 to 17.7] | 9.6 [2.6 to 16.7]

2. Secondary Outcome: Change in Reachable Workspace (RW) at 6 Months Post-Treatment
Description: Reachable Workspace (RW) is the area (cm^2) traced out when reaching for a target moving in a circular path just outside the reach of the participant.
Time Frame: 2 timepoints: prior to treatment, 6 months post-treatment
Measure: Least Squares Mean (95% Confidence Interval); unit: squared centimeters
Arm/Group | Arm+Hand CCFES | Hand CCFES | Arm+Hand Cyclic NMES
Number analyzed (Participants) | 21 | 24 | 8
squared centimeters | 430 [221 to 639] | 166 [55 to 276] | 152 [4 to 300]

3. Secondary Outcome: Change in Upper Extremity Fugl-Meyer (UEFM) Score at 6 Months Post-Treatment
Description: The Upper Extremity Fugl-Meyer (UEFM) is an assessment of motor impairment of the upper limb in which the participant is asked to make specific movements of the arm, forearm, wrist, and hand. Each movement is scored 0, 1, or 2 and the subscores are summed.
  Min=0; Max=66. Higher scores mean a better outcome.
Time Frame: 2 timepoints: prior to treatment, 6 months post-treatment
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Arm+Hand CCFES | Hand CCFES | Arm+Hand Cyclic NMES
Number analyzed (Participants) | 21 | 24 | 8
units on a scale | 11.0 [6.1 to 16.0] | 4.4 [0.9 to 7.9] | 10.7 [8.2 to 13.2]

4. Secondary Outcome: Change in Stroke Upper Limb Capacity Scale (SULCS) at 6 Months Post-Treatment
Description: Stroke Upper Limb Capacity Scale (SULCS) is a 10-item test in which participants are given a score of 0 or 1 on their performance of tasks requiring varying degrees of upper limb capacity.
  Min=0; Max=10. Higher scores mean a better outcome.
Time Frame: 2 timepoints: prior to treatment, 6 months post-treatment
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Arm+Hand CCFES | Hand CCFES | Arm+Hand Cyclic NMES
Number analyzed (Participants) | 21 | 24 | 8
units on a scale | 2.6 [1.2 to 3.9] | 1.5 [0.7 to 2.4] | 1.9 [1.1 to 2.8]

5. Secondary Outcome: Change in Arm Motor Abilities Test (AMAT) at 6 Months Post-Treatment
Description: The Arm Motor Abilities Test (AMAT) is an assessment of the participant's ability to do 9 standardized upper limb tasks. Each task is composed of 1 to 3 component tasks, each of which is rated on an ordinal scale of 0 to 5. The final score is the average of all component task scores across all 9 compound tasks.
  Min=0; Max=5. Higher scores mean a better outcome.
Time Frame: 2 timepoints: prior to treatment, 6 months post-treatment
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Arm+Hand CCFES | Hand CCFES | Arm+Hand Cyclic NMES
Number analyzed (Participants) | 21 | 24 | 8
units on a scale | 1.0 [0.5 to 1.6] | 0.8 [0.6 to 1.1] | 0.9 [0.5 to 1.4]

ADVERSE EVENTS:
Time Frame: From enrollment to 6-month post-treatment outcome assessment.
Arm/Group | Arm+Hand CCFES | Hand CCFES | Arm+Hand Cyclic NMES
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/28 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/28 | 0/11
Other Adverse Events (participants affected / at risk) | 4/28 | 7/28 | 2/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm+Hand CCFES (N=28) | Hand CCFES (N=28) | Arm+Hand Cyclic NMES (N=11)
Shoulder pain related to RW assessment (Musculoskeletal and connective tissue disorders) | 2 | 5 | 2
Numbness and Tingling in Both Hands (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Abdominal Pain During RW Assessment (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Transient Discomfort from Stimulation (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-02-01): https://cdn.clinicaltrials.gov/large-docs/56/NCT01688856/Prot_SAP_000.pdf